CLINICAL TRIAL: NCT02984371
Title: Ablation of the Epicardial Fat Pads to Treat Paroxysmal Atrial Fibrillation During Coronary Artery Bypass Grafting
Brief Title: Epicardial Fat Pads Ablation During Coronary Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASTR_0789
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Atrial Fibrillation; Ischemic Heart Disease
Keywords: atrial fibrillation; ganglionated plexi; ischemic heart disease
MeSH Terms: conditions — Atrial Fibrillation; Myocardial Ischemia | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Group 1 (Experimental): Coronary artery bypass grafting + epicardial ganglionated plexi ablation
  Interventions: Procedure: Coronary artery bypass grafting; Procedure: Epicardial ganglionated plexi ablation; Procedure: implantable loop recorder
- Group 2 (Active Comparator): Coronary artery bypass grafting
  Interventions: Procedure: Coronary artery bypass grafting; Procedure: implantable loop recorder

INTERVENTIONS:
Procedure: Coronary artery bypass grafting
Procedure: Epicardial ganglionated plexi ablation
  Arms: Group 1
Procedure: implantable loop recorder

SUMMARY:
The aim of this prospective randomized study was to assess the efficacy of ablation of the ganglionated plexi localized in the epicardial fat pads for preventing recurrences of atrial tachyarrhythmia in patients with paroxysmal atrial fibrillation undergoing coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* History of paroxysmal atrial fibrillation (recurrent episodes for at least 1 years, with 2 documented episodes over the last 6 months)
* Indication for cardiac surgery (e.g. coronary artery bypass grafting, valve repair/replacement) according to the American College of Cardiology/American Heart Association (ACC/AHA) guidelines for cardiac surgery

Exclusion Criteria:

Previous heart surgery or atrial fibrillation ablation procedure Emergency coronary artery bypass grafting Unstable angina or heart failure Persistent atrial fibrillation Planned maze procedure or pulmonary vein isolation Unwillingness to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence of any atrial tachyarrhythmia, including atrial fibrillation and atrial flutter/tachycardia, after cardiac surgery procedure with no antiarrhythmic drug | 12 month

SECONDARY OUTCOMES:
atrial fibrillation burden | 12 month
incidence of congestive heart failure | 12 month
incidence of sustained ventricular arrhythmias | 12 month
rehospitalization | 12 month
stroke or transient ischemic attack | 12 month
number of Deaths | 12 month

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - State Research Institute of CIrculation Pathology Novosibirsk, Russian Federation, Novosibirsk
  - Cardiology Research Institute, Tomsk